CLINICAL TRIAL: NCT00219089
Title: An Eight-week, Randomized, Double-blind, Parallel Group, Multicenter, Dose Escalation Study to Evaluate the Efficacy and Safety of Aliskiren Administered Alone and in Combination With Ramipril in Patients With Hypertension and Diabetes Mellitus
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of Aliskiren Alone and in Combination With Ramipril in Hypertensive, Diabetic Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2307
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Hypertension, Diabetes Mellitus
Keywords: Hypertension, aliskiren, blood pressure, diabetes mellitus, ramipril
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
To demonstrate the efficacy and safety of aliskiren given to patients with both hypertension and diabetes mellitus

ELIGIBILITY:
Inclusion Criteria

* Patients with essential hypertension
* Patients with a documented diagnosis of Type 1 or Type 2 diabetes mellitus.
* Patients who are eligible and able to participate in the study

Exclusion Criteria

* Severe hypertension
* History or evidence of a secondary form of hypertension
* History of hypertensive encephalopathy or cerebrovascular accident. Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2004-11; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting diastolic blood pressure after 8 weeks

SECONDARY OUTCOMES:
Change from baseline to week 4 endpoint in mean sitting diastolic blood pressure
Change from baseline to week 8 endpoint in mean sitting systolic blood pressure
Diastolic blood pressure less than 90 mmHg or reduction of 10 mmHg or greater from baseline after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Derived] Wang GM, Li LJ, Tang WL, Wright JM. Renin inhibitors versus angiotensin converting enzyme (ACE) inhibitors for primary hypertension. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD012569. doi: 10.1002/14651858.CD012569.pub2. PMID 33089502
- [Derived] Uresin Y, Taylor AA, Kilo C, Tschope D, Santonastaso M, Ibram G, Fang H, Satlin A. Efficacy and safety of the direct renin inhibitor aliskiren and ramipril alone or in combination in patients with diabetes and hypertension. J Renin Angiotensin Aldosterone Syst. 2007 Dec;8(4):190-8. doi: 10.3317/jraas.2007.028. PMID 18205098